CLINICAL TRIAL: NCT01428778
Title: Berlin Beat of Running Study - Frequency of Cardiac Arrhythmias & Cerebral Lesions in Marathon Runners
Brief Title: Berlin Beat of Running Study
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Center for Stroke Research Berlin (Other); Medical Institute BMW-Berlin Marathon, Berlin, Germany (Unknown)
Responsible Party: Principal Investigator, Karl Georg Haeusler, MD, Charite University, Berlin, Germany
Other Study IDs: Berlin Beat; EA4/042/11 (Other: Ethics Committee Charité - Universitätsmedizin Berlin)
Record Dates: First submitted 2011-08-31; First posted 2011-09-05 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Cardiac Arrhythmia; Brain Lesion; Stroke
Keywords: Marathon running; Brain MRI; ECG recording; Blood tests
MeSH Terms: conditions — Arrhythmias, Cardiac; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective observational study will investigate the frequency of new onset atrial fibrillation (AF) and of further cardiac arrhythmias as well as of (clinically silent) cerebral lesions in endurance runners before, during and after the BMW-Berlin Marathon 2011.

DETAILED DESCRIPTION:
Up to 120 experienced marathon runners will participate in the "Berlin Beat of Running Study" and will wear a transportable electrocardiogram (ECG) recorder at least 24 hours before, during and 24 hours after the BMW-Berlin Marathon. All participants will undergo brain MRI examinations to detect cerebral lesions within days before and after the marathon race, respectively. Moreover, serial blood samples will be taken a few days before, immediately after as well as a few days after the BMW-Berlin Marathon.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-65 years
* at least 2 marathon runs within the last 5 years
* weekly running of at least 40 km

Exclusion Criteria:

* Known cardiac arrhythmia or prior stroke
* contraindication for MRI.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experienced marathon runners
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Rate of cardiac arrhythmias in marathon runners detected by mobile ECG-recording | Up to 48 hours after the marathon race.
  During ECG recording

SECONDARY OUTCOMES:
Rate of (clinically silent) cerebral lesions detected by 3 Tesla brain MRI. | 3 days
  Up to 3 days after marathon.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Georg Haeusler, MD, Principal Investigator — Center for Stroke Research Berlin, Charité - Universitätsmedizin Berlin, Germany.; Matthias Endres, MD, Study Chair — Center for Stroke Research Berlin, Charité - Universitätsmedizin Berlin, Germany; Wilhelm Haverkamp, MD, Study Chair — Departement of Cardiology, Campus Virchow, Charité - Universitätsmedizin Berlin, Germany; Matthias Kruell, MD, Study Chair — Medical Institute BMW-Berlin Marathon; Peter U Heuschmann, MD, Study Chair — Center for Stroke Research Berlin; Gerhard Jan Jungehuelsing, MD, Principal Investigator — Center for Stroke Research Berlin
Locations (1):
- Center for Stroke Research Berlin, Berlin, Germany

REFERENCES:
- [Derived] Herm J, Topper A, Wutzler A, Kunze C, Krull M, Brechtel L, Lock J, Fiebach JB, Heuschmann PU, Haverkamp W, Endres M, Jungehulsing GJ, Haeusler KG. Frequency of exercise-induced ST-T-segment deviations and cardiac arrhythmias in recreational endurance athletes during a marathon race: results of the prospective observational Berlin Beat of Running study. BMJ Open. 2017 Aug 3;7(8):e015798. doi: 10.1136/bmjopen-2016-015798. PMID 28775185
- [Derived] Haeusler KG, Herm J, Kunze C, Krull M, Brechtel L, Lock J, Hohenhaus M, Heuschmann PU, Fiebach JB, Haverkamp W, Endres M, Jungehulsing GJ. Rate of cardiac arrhythmias and silent brain lesions in experienced marathon runners: rationale, design and baseline data of the Berlin Beat of Running study. BMC Cardiovasc Disord. 2012 Aug 31;12:69. doi: 10.1186/1471-2261-12-69. PMID 22938148